CLINICAL TRIAL: NCT02625090
Title: An Open-label, Multicenter, Extension Study to Evaluate the Long-term Safety, Tolerability, and Efficacy of UCB0942 When Used as Adjunctive Therapy for Partial-onset Seizures in Adult Subjects With Highly Drug-resistant Focal Epilepsy
Brief Title: An Open-label Extension Study of UCB0942 in Adult Patients With Highly Drug-resistant Focal Epilepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on available data, UCB has decided to stop development of padsevonil as adjunctive treatment of focal-onset seizure
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0073; 2015-001268-20 (EudraCT Number)
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Results first posted 2022-01-31 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Highly Drug-resistant Focal Epilepsy
Keywords: Drug-resistance; focal epilepsy; partial-onset seizures
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UCB0942 (Experimental): UCB0942 400 mg bid or a tapered UCB0942 dose of 200 mg bid.
  The Investigator will be allowed to increase or decrease the dose of UCB0942 to optimize tolerability and seizure control for each subject. Increases or decreases to the dose of UCB0942 should be made in steps not exceeding 200 mg/day per week; an exception is Taper Week 1 where a step of 800 mg/day to 500 mg/day is allowed. A faster decrease of the dose than 200 mg/day per week is allowed when it is clinically appropriate in the Investigator's medical judgment. Daily UCB0942 doses during this study may be 100 mg (50 mg bid), 200 mg (100 mg bid), 400 mg (200 mg bid), 600 mg (300 mg bid), or 800 mg (400 mg bid); intermediate doses will not be allowed except for tapering and titration unless agreed by the UCB Study Physician or PRA Medical Monitor. The dose of UCB0942 must always be administered as bid morning and evening doses, approximately 12 hours apart.
  Interventions: Drug: UCB0942

INTERVENTIONS:
Drug: UCB0942 — * Active Substance: UCB0942
  * Pharmaceutical form: Film-coated tablet
  * Concentration: 25 mg, 100 mg or 200 mg
  * Route of Administration: oral

SUMMARY:
The purpose of study EP0073 is to assess the long-term safety, tolerability, and efficacy during 5 years of treatment with the drug UCB0942 in patients with highly drug-resistant focal epilepsy. Also, the effects of UCB0942 on the patient's quality of life will be explored.

DETAILED DESCRIPTION:
For those subjects who benefit substantially from UCB0942 in the multicenter, randomized, double-blind, placebo-controlled, parallel group study EP0069, the current open-label extension study EP0073 will provide an opportunity to continue UCB0942 treatment after a careful evaluation of the individual benefit-risk balance and with close monitoring of safety, tolerability and efficacy of long-term study treatment.

ELIGIBILITY:
Inclusion Criteria:

* A written Informed Consent form approved by the Independent Ethics Committee is signed and dated by the subject, after the Investigator assesses whether the subject is able to understand the potential risks and benefits of participating in the study
* Subject must have completed Visit 13 (V13) of the Outpatient Maintenance Period of EP0069 to be eligible for enrollment into EP0073
* In EP0069, the subject demonstrated a reduction in frequency and/or severity of seizures as compared to baseline that is considered clinically significant by the Investigator and significant by the subject
* In EP0069, the subject experiences substantial benefit from UCB0942 with acceptable tolerability according to the subject and Investigator
* No tolerability issues that can outweigh attained benefits, in the opinion of the Investigator
* Female subjects of nonchildbearing potential (premenarcheal, postmenopausal for at least 2 years, bilateral oophorectomy or tubal ligation, and complete hysterectomy) are eligible. Female subjects of childbearing potential are eligible if they use medically accepted contraceptive methods
* Male subject confirms that, during the study period and for a period of 3 months after the final dose, when having sexual intercourse with a woman of childbearing potential, he will use a barrier contraceptive (eg, condom)Exclusion Criteria:
* Subject has active suicidal ideation as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the 'Since Last Visit' version of the Columbia Suicide Severity Rating Scale. The subject should be referred immediately to a Mental Healthcare Professional and must be withdrawn from the study
* Subject has taken other (non-Anti-Epileptic Drug) prescription, non-prescription, dietary (eg, grapefruit or passion fruit), or herbal products that are potent inducers or inhibitors of the CYP3A4 pathway for 2 weeks (or 5 half lives whichever is longer) prior to study entry
* Subject has an abnormality in the 12-lead electrocardiography that, in the opinion of the Investigator, increases the risks associated with participating in the study. In addition, any subject with any of the following findings will be excluded:

  1. Prolonged QTc (Bazett's, machine-read) interval defined as > 450 ms for males and > 470 ms for females
  2. Bundle branch blocks and other conduction abnormalities other than mild first degree atrioventricular block (defined as PR interval >= 220 ms)
  3. Irregular rhythms other than sinus arrhythmia or occasional, rare supraventricular or rare ventricular ectopic beats
  4. In the judgment of the Investigator, T-wave configurations are not of sufficient quality for assessing QT interval duration
* Subject has a clinically significant abnormality on echocardiography at the Entry Visit (V2) of EP0073
* Upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >ULN total bilirubin (>=1.5xULN total bilirubin if known Gilbert's syndrome) at the EV (V2) of EP0073 (V15 of EP0069). If subject has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (ie, direct bilirubin <35%). For enrolled subjects with a baseline result

  * ULN for ALT, AST, ALP, or total bilirubin, a baseline diagnosis and/or the cause of any clinically meaningful elevation must be understood and recorded in the electronic Case Report form (eCRF). If subject has >ULN ALT, AST, or ALP that does not meet the exclusion limit at screening (ie, the value is
  * ULN but <=2xULN at the EV [V2] of EP0073), repeat the tests, if possible, prior to dosing to ensure there is no further ongoing clinically relevant increase. In case of a clinically relevant increase, inclusion of the subject must be discussed with the Medical Monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (15):
- Belgium (3):
  - Ep0073 103, Brussels
  - Ep0073 101, Ghent
  - Ep0073 102, Leuven
- Ep0073 201, Sofia, Bulgaria
- Germany (3):
  - Ep0073 402, Bielefeld
  - Ep0073 403, Radeberg
  - Ep0073 405, Ravensburg
- Hungary (2):
  - Ep0073 601, Budapest
  - Ep0073 602, Budapest
- Ep0073 302, Heeze, Netherlands
- Spain (5):
  - Ep0073 502, Barcelona
  - Ep0073 505, L'Hospitalet de Llobregat
  - Ep0073 506, Madrid
  - Ep0073 501, Seville
  - Ep0073 503, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in December 2015 and concluded in November 2020.
Pre-assignment Details: Participant flow refers to the Safety Set. Participants who experienced substantial benefit from UCB0942 with acceptable tolerability in the EP0069 (NCT02495844) study had opportunity to continue treatment in this study.
Groups:
- UCB0942: All enrolled participants continued the same UCB0942 dose which they were receiving during last visit of study EP0069 and the dose could be further increased or decreased in participants to optimize the drug tolerability and seizure control for each participant. Daily UCB0942 film-coated tablets were administered orally in doses of 100 milligrams (mg) (50 mg twice daily [bid]), 200 mg (100 mg bid), 400 mg (200 mg bid), 600 mg (300 mg bid), or 800 mg (400 mg bid) for up to approximately 5 years.
Period: Overall Study
Arm/Group | UCB0942
Started | 42
Completed | 0
Not Completed | 42
Not completed — Participant wants to be pregnant | 2
Not completed — For the Promoter | 1
Not completed — Sponsor's Decision | 9
Not completed — Somnolence | 1
Not completed — Study terminated by Sponsor | 7
Not completed — Negative Benefit/Risk | 1
Not completed — Protocol Deviation | 2
Not completed — Lack of Efficacy | 16
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) consisted of all enrolled study participants who took at least 1 dose of UCB0942 in the EP0073 study.
Groups:
- UCB0942: All enrolled participants continued the same UCB0942 dose which they were receiving during last visit of study EP0069 and the dose could be further increased or decreased in participants to optimize the drug tolerability and seizure control for each participant. Daily UCB0942 film-coated tablets were administered orally in doses of 100 mg (50 mg twice daily [bid]), 200 mg (100 mg bid), 400 mg (200 mg bid), 600 mg (300 mg bid), or 800 mg (400 mg bid) for up to approximately 5 years.
Arm/Group | UCB0942
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40
  Other/mixed | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing at Least One Treatment-Emergent Adverse Event (TEAE) From the Beginning at Entry Visit (EV) of the Evaluation Period to End of Safety Follow-Up Visit During the EP0073 Study
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
  Percentage of participants experiencing at least one treatment-emergent adverse event (reported by the participant and/or caregiver or observed by the Investigator or inpatient staff) are reported.
Time Frame: From Entry Visit to End of Safety Follow-Up Visit (up to 5 years)
Population: The Safety Set (SS) consisted of all enrolled study participants who took at least 1 dose of UCB0942 in the EP0073 study.
Measure: Number; unit: percentage of participants
Groups:
- UCB0942 (SS): All enrolled participants continued the same UCB0942 dose which they were receiving during last visit of study EP0069 and the dose could be further increased or decreased in participants to optimize the drug tolerability and seizure control for each participant. Daily UCB0942 film-coated tablets were administered orally in doses of 100 mg (50 mg bid), 200 mg (100 mg bid), 400 mg (200 mg bid), 600 mg (300 mg bid), or 800 mg (400 mg bid) for up to approximately 5 years. Participants formed the Safety Set (SS).
Arm/Group | UCB0942 (SS)
Number analyzed (Participants) | 42
percentage of participants | 90.5

2. Primary Outcome: 75% Responder Rate by 3-month Interval (Month 0 to 3) Over the Evaluation Period
Description: A 75% responder is defined as a participant with a ≥75% reduction in partial-onset seizure (POS) frequency for observable focal-onset seizures relative to the 2-week Prospective Outpatient Baseline Period defined in EP0069. Observable focal-onset seizures refer to Type IA1 (simple partial seizures with motor signs), IB (complex partial seizures), and IC (partial seizures evolving to secondarily generalized seizures) of the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures, 1981. It was calculated using formula: Count of 75% responders during the Period/ number of participants during the Period × 100.
Time Frame: Over 3-month interval over the Evaluation Period (Month 0-3)
Population: The Full Analysis Set (FAS) consisted of all enrolled study participants who took at least 1 dose of UCB0942 and completed at least 1 seizure diary during the Evaluation Period in EP0073. Here, number of participants analyzed included those participants who were evaluable for the assessment.
Measure: Number; unit: percentage of participants
Groups:
- UCB0942 (FAS): All enrolled participants continued the same UCB0942 dose which they were receiving during last visit of study EP0069 and the dose could be further increased or decreased in participants to optimize the drug tolerability and seizure control for each participant. Daily UCB0942 film-coated tablets were administered orally in doses of 100 mg (50 mg bid), 200 mg (100 mg bid), 400 mg (200 mg bid), 600 mg (300 mg bid), or 800 mg (400 mg bid) for up to approximately 5 years. Participants formed the FAS.
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 41
percentage of participants | 24.4

3. Secondary Outcome: Median Partial-onset Seizure Frequency Per 28 Days by 3-month Intervals Over the Evaluation Period of the EP0073 Study
Description: Median partial-onset seizure frequency per 28 days by 3-month intervals over the Evaluation Period of the EP0073 study was reported.
Time Frame: Over the 3-month interval: Month 0-3, >3-6, >6-9, >9-12, >12-15, >15-18, >18-21, >21-24, >24-27, >27-30, >30-33, >33-36, >36-39, >39-42, >42-45, >45-48, >48-51, >51-54, >54-57 over the Evaluation Period
Population: The FAS consisted of all enrolled study participants who took at least 1 dose of UCB0942 and completed at least 1 seizure diary during the Evaluation Period in EP0073. Here, number analyzed signifies participants who were evaluable at specified time points.
Measure: Median (Inter-Quartile Range); unit: seizure frequency per 28 days
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 42
seizure frequency per 28 days
  Month 0-3 | 18.98 [10.89 to 48.22]
  Month >3-6 | 22.99 [13.07 to 66.18]
  Month >6-9: number analyzed (Participants) | 35
  Month >6-9 | 23.33 [8.09 to 56.00]
  Month >9-12: number analyzed (Participants) | 29
  Month >9-12 | 18.67 [6.84 to 37.96]
  Month >12-15: number analyzed (Participants) | 27
  Month >12-15 | 23.23 [9.02 to 49.47]
  Month >15-18: number analyzed (Participants) | 27
  Month >15-18 | 19.91 [11.20 to 41.48]
  Month >18-21: number analyzed (Participants) | 27
  Month >18-21 | 16.80 [8.09 to 42.00]
  Month >21-24: number analyzed (Participants) | 23
  Month >21-24 | 14.31 [5.91 to 36.09]
  Month >24-27: number analyzed (Participants) | 24
  Month >24-27 | 14.31 [8.71 to 38.53]
  Month >27-30: number analyzed (Participants) | 22
  Month >27-30 | 14.16 [5.91 to 38.58]
  Month >30-33: number analyzed (Participants) | 21
  Month >30-33 | 16.80 [7.78 to 42.62]
  Month >33-36: number analyzed (Participants) | 21
  Month >33-36 | 19.29 [6.84 to 46.67]
  Month >36-39: number analyzed (Participants) | 19
  Month >36-39 | 13.69 [7.16 to 45.11]
  Month >39-42: number analyzed (Participants) | 19
  Month >39-42 | 9.96 [5.91 to 57.24]
  Month >42-45: number analyzed (Participants) | 15
  Month >42-45 | 13.07 [3.73 to 63.17]
  Month >45-48: number analyzed (Participants) | 11
  Month >45-48 | 10.58 [2.80 to 59.42]
  Month >48-51: number analyzed (Participants) | 11
  Month >48-51 | 9.02 [1.56 to 48.16]
  Month >51-54: number analyzed (Participants) | 6
  Month >51-54 | 7.80 [3.73 to 33.60]
  Month >54-57: number analyzed (Participants) | 1
  Month >54-57 | 7.84 [7.84 to 7.84]

4. Secondary Outcome: Median Partial-onset Seizure Frequency Per 28 Days by Seizure Type by 3-month Intervals Over the Evaluation Period of the EP0073 Study
Description: Median partial-onset seizure frequency per 28 days by seizure type (Type IA1, Type IB, Type IC) by 3-month intervals over the Evaluation Period of the EP0073 study was reported. Observable focal-onset seizures refer to Type IA1 (simple partial seizures with motor signs), IB (complex partial seizures), and IC (partial seizures evolving to secondarily generalized seizures) of the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures, 1981.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: seizure frequency per 28 days
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 42
seizure frequency per 28 days
  Type IA1: Month 0-3 | 0.00 [0.00 to 2.18]
  Type IA1: Month >3-6 | 0.00 [0.00 to 7.47]
  Type IA1: Month >6-9: number analyzed (Participants) | 35
  Type IA1: Month >6-9 | 0.00 [0.00 to 4.36]
  Type IA1: Month >9-12: number analyzed (Participants) | 29
  Type IA1: Month >9-12 | 0.00 [0.00 to 0.00]
  Type IA1: Month >12-15: number analyzed (Participants) | 27
  Type IA1: Month >12-15 | 0.00 [0.00 to 1.24]
  Type IA1: Month >15-18: number analyzed (Participants) | 27
  Type IA1: Month >15-18 | 0.00 [0.00 to 1.87]
  Type IA1: Month >18-21: number analyzed (Participants) | 27
  Type IA1: Month >18-21 | 0.00 [0.00 to 4.36]
  Type IA1: Month >21-24: number analyzed (Participants) | 23
  Type IA1: Month >21-24 | 0.00 [0.00 to 2.80]
  Type IA1: Month >24-27: number analyzed (Participants) | 24
  Type IA1: Month >24-27 | 0.00 [0.00 to 3.27]
  Type IA1: Month >27-30: number analyzed (Participants) | 22
  Type IA1: Month >27-30 | 0.00 [0.00 to 0.93]
  Type IA1: Month >30-33: number analyzed (Participants) | 21
  Type IA1: Month >30-33 | 0.00 [0.00 to 2.49]
  Type IA1: Month >33-36: number analyzed (Participants) | 21
  Type IA1: Month >33-36 | 0.00 [0.00 to 2.49]
  Type IA1: Month >36-39: number analyzed (Participants) | 19
  Type IA1: Month >36-39 | 0.00 [0.00 to 3.42]
  Type IA1: Month >39-42: number analyzed (Participants) | 19
  Type IA1: Month >39-42 | 0.00 [0.00 to 2.80]
  Type IA1: Month >42-45: number analyzed (Participants) | 15
  Type IA1: Month >42-45 | 0.00 [0.00 to 7.47]
  Type IA1: Month >45-48: number analyzed (Participants) | 11
  Type IA1: Month >45-48 | 0.00 [0.00 to 4.67]
  Type IA1: Month >48-51: number analyzed (Participants) | 11
  Type IA1: Month >48-51 | 0.00 [0.00 to 3.73]
  Type IA1: Month >51-54: number analyzed (Participants) | 6
  Type IA1: Month >51-54 | 0.00 [0.00 to 1.87]
  Type IA1: Month >54-57: number analyzed (Participants) | 1
  Type IA1: Month >54-57 | 4.48 [4.48 to 4.48]
  Type IB: Month 0-3 | 10.73 [4.67 to 35.00]
  Type IB: Month >3-6 | 12.67 [1.56 to 28.00]
  Type IB: Month >6-9: number analyzed (Participants) | 35
  Type IB: Month >6-9 | 9.33 [0.00 to 34.68]
  Type IB: Month >9-12: number analyzed (Participants) | 29
  Type IB: Month >9-12 | 9.64 [1.24 to 26.11]
  Type IB: Month >12-15: number analyzed (Participants) | 27
  Type IB: Month >12-15 | 15.56 [0.93 to 34.84]
  Type IB: Month >15-18: number analyzed (Participants) | 27
  Type IB: Month >15-18 | 13.38 [2.18 to 37.64]
  Type IB: Month >18-21: number analyzed (Participants) | 27
  Type IB: Month >18-21 | 13.07 [0.62 to 33.91]
  Type IB: Month >21-24: number analyzed (Participants) | 23
  Type IB: Month >21-24 | 7.78 [0.93 to 25.20]
  Type IB: Month >24-27: number analyzed (Participants) | 24
  Type IB: Month >24-27 | 9.80 [2.49 to 27.38]
  Type IB: Month >27-30: number analyzed (Participants) | 22
  Type IB: Month >27-30 | 9.49 [1.87 to 33.75]
  Type IB: Month >30-33: number analyzed (Participants) | 21
  Type IB: Month >30-33 | 9.64 [3.11 to 32.98]
  Type IB: Month >33-36: number analyzed (Participants) | 21
  Type IB: Month >33-36 | 7.47 [2.49 to 25.67]
  Type IB: Month >36-39: number analyzed (Participants) | 19
  Type IB: Month >36-39 | 6.53 [3.73 to 35.47]
  Type IB: Month >39-42: number analyzed (Participants) | 19
  Type IB: Month >39-42 | 6.84 [0.31 to 24.58]
  Type IB: Month >42-45: number analyzed (Participants) | 15
  Type IB: Month >42-45 | 5.29 [2.18 to 20.84]
  Type IB: Month >45-48: number analyzed (Participants) | 11
  Type IB: Month >45-48 | 4.36 [1.24 to 26.96]
  Type IB: Month >48-51: number analyzed (Participants) | 11
  Type IB: Month >48-51 | 4.67 [0.31 to 43.87]
  Type IB: Month >51-54: number analyzed (Participants) | 6
  Type IB: Month >51-54 | 3.29 [1.06 to 33.60]
  Type IB: Month >54-57: number analyzed (Participants) | 1
  Type IB: Month >54-57 | 3.36 [3.36 to 3.36]
  Type IC: Month 0-3 | 0.00 [0.00 to 0.00]
  Type IC: Month >3-6 | 0.00 [0.00 to 0.00]
  Type IC: Month >6-9: number analyzed (Participants) | 35
  Type IC: Month >6-9 | 0.00 [0.00 to 0.00]
  Type IC: Month >9-12: number analyzed (Participants) | 29
  Type IC: Month >9-12 | 0.00 [0.00 to 0.00]
  Type IC: Month >12-15: number analyzed (Participants) | 27
  Type IC: Month >12-15 | 0.00 [0.00 to 0.00]
  Type IC: Month >15-18: number analyzed (Participants) | 27
  Type IC: Month >15-18 | 0.00 [0.00 to 0.00]
  Type IC: Month >18-21: number analyzed (Participants) | 27
  Type IC: Month >18-21 | 0.00 [0.00 to 0.00]
  Type IC: Month >21-24: number analyzed (Participants) | 23
  Type IC: Month >21-24 | 0.00 [0.00 to 0.00]
  Type IC: Month >24-27: number analyzed (Participants) | 24
  Type IC: Month >24-27 | 0.00 [0.00 to 0.00]
  Type IC: Month >27-30: number analyzed (Participants) | 22
  Type IC: Month >27-30 | 0.00 [0.00 to 0.00]
  Type IC: Month >30-33: number analyzed (Participants) | 21
  Type IC: Month >30-33 | 0.00 [0.00 to 0.00]
  Type IC: Month >33-36: number analyzed (Participants) | 21
  Type IC: Month >33-36 | 0.00 [0.00 to 0.00]
  Type IC: Month >36-39: number analyzed (Participants) | 19
  Type IC: Month >36-39 | 0.00 [0.00 to 0.31]
  Type IC: Month >39-42: number analyzed (Participants) | 19
  Type IC: Month >39-42 | 0.00 [0.00 to 0.00]
  Type IC: Month >42-45: number analyzed (Participants) | 15
  Type IC: Month >42-45 | 0.00 [0.00 to 0.00]
  Type IC: Month >45-48: number analyzed (Participants) | 11
  Type IC: Month >45-48 | 0.00 [0.00 to 0.31]
  Type IC: Month >48-51: number analyzed (Participants) | 11
  Type IC: Month >48-51 | 0.00 [0.00 to 0.31]
  Type IC: Month >51-54: number analyzed (Participants) | 6
  Type IC: Month >51-54 | 0.00 [0.00 to 1.87]
  Type IC: Month >54-57: number analyzed (Participants) | 1
  Type IC: Month >54-57 | 0.00 [0.00 to 0.00]

5. Secondary Outcome: Percent Change in Partial-onset Seizure Frequency Relative to the Baseline Period Defined in EP0069 by 3-month Intervals Over the Evaluation Period of the EP0073 Study
Description: Percent change from Baseline in seizure frequency for observable focal-onset seizures (Type IA1, IB, and IC) to the corresponding interval was calculated using the following formula: change from Baseline in the 28 day adjusted seizure frequency/28 day adjusted seizure frequency during the EP0069 2- week Prospective Outpatient Baseline Period × 100. The numerator is calculated by subtracting the 28-day adjusted seizure frequency during the Period of interest from the 28-day adjusted seizure frequency during the EP0069 2-week prospective outpatient Baseline Period. Observable focal-onset seizures refer to Type IA1 (simple partial seizures with motor signs), IB (complex partial seizures), and IC (partial seizures evolving to secondarily generalized seizures) of the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures, 1981.
Time Frame: Over the 3-month interval: Month 0-3, >3-6, >6-9, >9-12, >12-15, >15-18, >18-21, >21-24, >24-27, >27-30, >30-33, >33-36, >36-39, >39-42, >42-45, >45-48, >48-51, >51-54, >54-57 over the Evaluation Period, Relative to Baseline (of EP0069)
Population: The FAS consisted of all enrolled study participants who took at least 1 dose of UCB0942 and completed at least 1 seizure diary during the Evaluation Period in EP0073. Here, number of participants analyzed included those participants who were evaluable for the assessment and number analyzed signifies participants who were evaluable at specified time points.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 41
percent change
  Month 0-3 | 50.51 [21.74 to 72.53]
  Month >3-6 | 39.14 [12.50 to 72.78]
  Month >6-9: number analyzed (Participants) | 34
  Month >6-9 | 56.98 [31.19 to 72.22]
  Month >9-12: number analyzed (Participants) | 28
  Month >9-12 | 62.22 [39.99 to 80.54]
  Month >12-15: number analyzed (Participants) | 26
  Month >12-15 | 55.74 [40.95 to 72.78]
  Month >15-18: number analyzed (Participants) | 26
  Month >15-18 | 54.04 [35.71 to 72.72]
  Month >18-21: number analyzed (Participants) | 26
  Month >18-21 | 57.27 [39.42 to 76.28]
  Month >21-24: number analyzed (Participants) | 22
  Month >21-24 | 68.57 [46.67 to 76.67]
  Month >24-27: number analyzed (Participants) | 23
  Month >24-27 | 60.15 [40.31 to 77.41]
  Month >27-30: number analyzed (Participants) | 21
  Month >27-30 | 59.82 [44.79 to 80.06]
  Month >30-33: number analyzed (Participants) | 20
  Month >30-33 | 59.57 [41.94 to 76.17]
  Month >33-36: number analyzed (Participants) | 20
  Month >33-36 | 59.73 [35.42 to 78.96]
  Month >36-39: number analyzed (Participants) | 18
  Month >36-39 | 64.50 [45.56 to 78.90]
  Month >39-42: number analyzed (Participants) | 18
  Month >39-42 | 59.01 [37.78 to 80.06]
  Month >42-45: number analyzed (Participants) | 14
  Month >42-45 | 68.79 [38.39 to 80.00]
  Month >45-48: number analyzed (Participants) | 10
  Month >45-48 | 68.17 [56.98 to 85.00]
  Month >48-51: number analyzed (Participants) | 10
  Month >48-51 | 67.12 [51.67 to 91.67]
  Month >51-54: number analyzed (Participants) | 5
  Month >51-54 | 73.08 [61.92 to 80.00]
  Month >54-57: number analyzed (Participants) | 1
  Month >54-57 | 73.56 [73.56 to 73.56]

6. Secondary Outcome: 50% Responder Rate by 3-month Intervals Over the Evaluation Period of the EP0073 Study
Description: A 50% responder was defined as a participant with a ≥50% reduction in partial-onset seizure (POS) frequency for observable focal-onset seizures relative to the 2-week Prospective Outpatient Baseline Period defined in EP0069. Observable focal-onset seizures refer to Type IA1 (simple partial seizures with motor signs), IB (complex partial seizures), and IC (partial seizures evolving to secondarily generalized seizures) of the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures, 1981. It was calculated using formula: Count of 50% responders during the period/number of participants during the period × 100.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 41
percentage of participants
  Month 0-3 | 51.2
  Month >3-6 | 39.0
  Month >6-9: number analyzed (Participants) | 34
  Month >6-9 | 58.8
  Month >9-12: number analyzed (Participants) | 28
  Month >9-12 | 67.9
  Month >12-15: number analyzed (Participants) | 26
  Month >12-15 | 65.4
  Month >15-18: number analyzed (Participants) | 26
  Month >15-18 | 53.8
  Month >18-21: number analyzed (Participants) | 26
  Month >18-21 | 57.7
  Month >21-24: number analyzed (Participants) | 22
  Month >21-24 | 72.7
  Month >24-27: number analyzed (Participants) | 23
  Month >24-27 | 69.6
  Month >27-30: number analyzed (Participants) | 21
  Month >27-30 | 66.7
  Month >30-33: number analyzed (Participants) | 20
  Month >30-33 | 70.0
  Month >33-36: number analyzed (Participants) | 20
  Month >33-36 | 65.0
  Month >36-39: number analyzed (Participants) | 18
  Month >36-39 | 72.2
  Month >39-42: number analyzed (Participants) | 18
  Month >39-42 | 72.2
  Month >42-45: number analyzed (Participants) | 14
  Month >42-45 | 64.3
  Month >45-48: number analyzed (Participants) | 10
  Month >45-48 | 80.0
  Month >48-51: number analyzed (Participants) | 10
  Month >48-51 | 90.0
  Month >51-54: number analyzed (Participants) | 5
  Month >51-54 | 80.0
  Month >54-57: number analyzed (Participants) | 1
  Month >54-57 | 100

7. Secondary Outcome: Percentage of Seizure-free Days by 3-month Intervals Over the Evaluation Period
Description: The number of seizure-free days is defined as the total number of days within an analysis Period or time interval for which no seizures were reported. The percentage of seizure-free days is to be computed as 100 times the number of seizure-free days divided by the number of days for which daily diary data was available in the specified analysis Period. Days without the corresponding daily diary data (ie, "Not Done" is ticked) are not used in these computations.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: percentage of days
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 42
percentage of days
  Month 0-3 | 48.33 [24.44 to 76.67]
  Month >3-6 | 42.81 [8.89 to 68.89]
  Month >6-9: number analyzed (Participants) | 35
  Month >6-9 | 54.44 [10.00 to 80.00]
  Month >9-12: number analyzed (Participants) | 29
  Month >9-12 | 55.56 [25.56 to 78.89]
  Month >12-15: number analyzed (Participants) | 27
  Month >12-15 | 54.44 [22.22 to 78.89]
  Month >15-18: number analyzed (Participants) | 27
  Month >15-18 | 51.11 [25.56 to 73.33]
  Month >18-21: number analyzed (Participants) | 27
  Month >18-21 | 61.11 [26.67 to 80.00]
  Month >21-24: number analyzed (Participants) | 23
  Month >21-24 | 57.78 [30.00 to 86.67]
  Month >24-27: number analyzed (Participants) | 24
  Month >24-27 | 60.00 [31.11 to 77.22]
  Month >27-30: number analyzed (Participants) | 22
  Month >27-30 | 64.44 [22.22 to 85.56]
  Month >30-33: number analyzed (Participants) | 21
  Month >30-33 | 57.78 [28.89 to 80.00]
  Month >33-36: number analyzed (Participants) | 21
  Month >33-36 | 60.00 [21.11 to 77.78]
  Month >36-39: number analyzed (Participants) | 19
  Month >36-39 | 68.89 [24.44 to 77.78]
  Month >39-42: number analyzed (Participants) | 19
  Month >39-42 | 67.78 [16.67 to 88.89]
  Month >42-45: number analyzed (Participants) | 15
  Month >42-45 | 67.78 [6.67 to 86.67]
  Month >45-48: number analyzed (Participants) | 11
  Month >45-48 | 72.22 [11.11 to 91.11]
  Month >48-51: number analyzed (Participants) | 11
  Month >48-51 | 73.33 [4.00 to 94.44]
  Month >51-54: number analyzed (Participants) | 6
  Month >51-54 | 80.65 [6.06 to 86.67]
  Month >54-57: number analyzed (Participants) | 1
  Month >54-57 | 72.00 [72.00 to 72.00]

8. Secondary Outcome: Seizure-free Rate Over the Evaluation Period
Description: Participants were considered seizure free for a given Period or time interval if the participant, completes the Period or time interval, reports no seizures during the Period, and has no more than 10% of days in the Period for which seizure data is not available (ie, "Not Done" is reported on the Seizure Count CRF). The seizure freedom rate (%) for a specific time Period was calculated using the following formula: Count of seizure free participants during the Period/ Number of participants during the Period × 100.
Time Frame: Over the Evaluation Period (up to 5 years)
Population: The FAS consisted of all enrolled study participants who took at least 1 dose of UCB0942 and completed at least 1 seizure diary during the Evaluation Period in EP0073.
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 42
percentage of participants | 0

9. Secondary Outcome: Changes in Quality of Life in Epilepsy 31-P (QOLIE-31-P) Total Score From Visit 3 (Week 2) of EP0069 Through the Assessment of the Evaluation Period of EP0073
Description: The QOLIE-31-P includes 30 items grouped into 7 multi-item subscales (seizure worry, overall quality of life, emotional well-being, energy/fatigue, cognitive functioning, medication effects, and social function) and a health status item. Individual responses for the 30 subscale items are rescaled to 0 to 100 with higher scores reflecting better functioning. Each subscale score is then calculated by summing rescaled responses for that subscale and dividing by number of items with non-missing response. Responses for health status item are multiple of 10 ranging from 0 to 100 with a higher score corresponding to better health status. The QOLIE-31-P total score was calculated as weighted sum of the subscale scores which ranges from 0 to 100 with higher score reflecting better functioning.
Time Frame: Month 3, 7, 13, 19, 25, 31, 37, 43, 49, early discontinuation visit (EDV) (up to Month 58), Relative to Baseline (of EP0069)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 39
scores on a scale
  Month 3 | 3.1 (14.2)
  Month 7: number analyzed (Participants) | 31
  Month 7 | 3.8 (17.0)
  Month 13: number analyzed (Participants) | 25
  Month 13 | 6.8 (17.7)
  Month 19: number analyzed (Participants) | 24
  Month 19 | 5.7 (18.0)
  Month 25: number analyzed (Participants) | 22
  Month 25 | 4.7 (24.8)
  Month 31: number analyzed (Participants) | 20
  Month 31 | 5.4 (21.7)
  Month 37: number analyzed (Participants) | 18
  Month 37 | 3.4 (18.8)
  Month 43: number analyzed (Participants) | 13
  Month 43 | 1.0 (19.0)
  Month 49: number analyzed (Participants) | 4
  Month 49 | -4.6 (22.2)
  EDV (up to Month 58): number analyzed (Participants) | 38
  EDV (up to Month 58) | 2.2 (19.9)

10. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >3-6) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >3-6)
Population: The FAS consisted of all enrolled study participants who took at least 1 dose of UCB0942 and completed at least 1 seizure diary during the Evaluation Period in EP0073. Here, number of participants analyzed included those participants who were evaluable for the assessment.
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 41
percentage of participants | 24.4

11. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >6-9) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >6-9)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 34
percentage of participants | 20.6

12. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >9-12) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >9-12)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 28
percentage of participants | 28.6

13. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >12-15) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >12-15)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 26
percentage of participants | 23.1

14. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >15-18) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >15-18)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 26
percentage of participants | 23.1

15. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >18-21) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >18-21)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 26
percentage of participants | 26.9

16. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >21-24) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >21-24)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 22
percentage of participants | 27.3

17. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >24-27) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >24-27)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 23
percentage of participants | 26.1

18. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >27-30) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >27-30)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 21
percentage of participants | 33.3

19. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >30-33) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >30-33)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 20
percentage of participants | 25.0

20. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >33-36) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >33-36)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 20
percentage of participants | 35.0

21. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >36-39) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >36-39)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 18
percentage of participants | 27.8

22. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >39-42) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >39-42)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 18
percentage of participants | 27.8

23. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >42-45) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >42-45)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 14
percentage of participants | 50.0

24. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >45-48) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >45-48)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 10
percentage of participants | 40.0

25. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >48-51) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >48-51)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 10
percentage of participants | 40.0

26. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >51-54) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >51-54)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 5
percentage of participants | 40.0

27. Primary Outcome: 75% Responder Rate by 3-month Interval (Month >54-57) Over the Evaluation Period
Description: as for outcome 2
Time Frame: Over 3-month interval over the Evaluation Period (Month >54-57)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | UCB0942 (FAS)
Number analyzed (Participants) | 1
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: From Entry Visit to End of Safety Follow-Up Visit (up to approximately 5 years)
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) that started on or after the first dose of UCB0942 in EP0073 or AEs whose intensity worsened on or after the date of first dose of UCB0942 in EP0073.
Arm/Group | UCB0942 (SS)
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 12/42
Other Adverse Events (participants affected / at risk) | 32/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UCB0942 (SS) (N=42)
Cellulitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2)
Seizure (Nervous system disorders) | 3 (3)
Status epilepticus (Nervous system disorders) | 2 (3)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Seizure cluster (Nervous system disorders) | 1 (1)
Myomectomy (Surgical and medical procedures) | 1 (1)
Therapy change (Surgical and medical procedures) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UCB0942 (SS) (N=42)
Vomiting (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 9 (13)
Nasopharyngitis (Infections and infestations) | 6 (9)
Gastroenteritis (Infections and infestations) | 4 (4)
Respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 4 (4)
Weight increased (Investigations) | 6 (6)
Somnolence (Nervous system disorders) | 11 (16)
Dizziness (Nervous system disorders) | 7 (8)
Headache (Nervous system disorders) | 6 (6)
Memory impairment (Nervous system disorders) | 4 (4)
Depressed mood (Psychiatric disorders) | 3 (5)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Irritability (Psychiatric disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT02625090/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT02625090/SAP_001.pdf